CLINICAL TRIAL: NCT03061253
Title: Impact on Cardiovascular Function in Smokers Making a Quit Attempt Using E-cigarettes Compared With Smokers Making a Quit Attempt With Prescription Nicotine-Replacement Therapy
Brief Title: E-cigarettes and Cardiovascular Function
Acronym: ISME-NRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: King's College London (Other); Heart Research U.K. (Unknown); Help2Change (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HWB-2016-17-S&E-10
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Smoking Cessation; Cardiovascular Diseases; Microcirculation; Macrocirculation
Keywords: Electronic Cigarettes; Laser Doppler Flowmetry; Ultrasound; Nicotine Replacement Therapy
MeSH Terms: conditions — Smoking Cessation; Cardiovascular Diseases; Vaping | interventions — Electronic Nicotine Delivery Systems; Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nicotine-inclusive e-cigarettes (Experimental): Participants will receive e-cigarettes (nicotine-inclusive) combined with behavioural change support over a 3 month period.
  Interventions: Other: Electronic Cigarette and behavioural change support.
- Nicotine-free e-cigarettes (Experimental): Participants will receive e-cigarettes (nicotine-free) combined with behavioural change support over a 3 month period.
  Interventions: Other: Nicotine-Free Electronic Cigarette and behavioural change support.
- Nicotine Replacement Therapy (NRT) (Active Comparator): Participants will be referred to smoking cessation services where they will be expected to receive Nicotine Replacement Therapy combined with behavioural change support over a 3 month period.
  Interventions: Other: Nicotine Replacement Therapy and behavioural change support.

INTERVENTIONS:
Other: Electronic Cigarette and behavioural change support. — The nicotine strength of Group A (nicotine-inclusive e-cigarettes) cartridges will be 18 mg/ml of nicotine strength. All participants will receive up to 6 behavioural change support sessions over the 3-month intervention period.
  Other Names: e-cigarette
  Arms: Nicotine-inclusive e-cigarettes
Other: Nicotine-Free Electronic Cigarette and behavioural change support. — Group B participants will receive nicotine-free cartridges for the period of the intervention. All participants will receive up to 6 behavioural change support sessions over the 3-month intervention period.
  Other Names: Nicotine-free e-cigarette
  Arms: Nicotine-free e-cigarettes
Other: Nicotine Replacement Therapy and behavioural change support. — Group C participants will be referred to smoking cessation services where they will be expected to receive Nicotine Replacement Therapy and up to 6 behavioural change support sessions over the 3-month intervention period, as per current guidelines.
  Other Names: NRT
  Arms: Nicotine Replacement Therapy (NRT)

SUMMARY:
The large current uptake of e-cigarettes (2.8 million U.K. users in 2016; 26), the continuous involvement of e-cigarettes (which potentially affects their contents as well), the uncertainty about their medium- and longer-term effects, and the need to promote smoking cessation as means of reducing Cardiovascular disease, dictate that more research is urgently needed. Research exploring the impact of e-cigarettes on cardiovascular function/ health has been requested by the European Parliament, the British Medical Association, regulatory agencies, clinicians and researchers, as there is currently no consensus within the smoking cessation community as to the potential impact of e-cigarettes. With e-cigarettes being successful in replacing traditional cigarettes (i.e. up to 42% within a month), such studies should not only be efficacy-focused, but should also explore the physiological effects of e-cigarettes, as preliminary work in the field is contrasting and limited, in both the acute- and longer-term timeframe. Furthermore, as e-cigarettes are not simple nicotine-based products, the general public, researchers and government agencies cannot rely on the existing research exploring the effects of nicotine on the cardio-vasculature (e.g. coronary and peripheral vasoconstriction, intravascular inflammation and deregulation of cardiac autonomic function as well as inhibition of microcirculation). Thus, the lack of direct evidence - which would clarify the degree of safety of e-cigarettes for the user's vascular system and determine their longer-term cardiovascular disease risk - increases the need for research in the field.

Such studies will supply in-depth information to service-users and policy-makers, especially as the recently-initiated U.K.'s "Medicines and Healthcare Products Regulatory Agency" validation of e-cigarettes will increase likelihood of their introduction in smoking cessation clinics.

This study will bridge the existing knowledge gap and inform the general public, the scientific and the smoking cessation community in respect to the physiological (e.g. cardiovascular health) and participants' experience of both nicotine-inclusive and nicotine-free, e-cigarettes (when combined with behavioural change support) and compare it against a currently NHS-applied smoking cessation pathway that combines Nicotine Replacement Therapy and behavioural change support. This will allow future research to advance and optimize the pharmacological treatment of tobacco and nicotine dependence, by taking into consideration the study's physiological and Health Economics' findings.

ELIGIBILITY:
Inclusion Criteria:

* smokers (at least 10 cigarettes/ day for the past year)
* willing to attempt quit smoking by using the National Health Service smoking cessation services or via e-cigarette use.

Exclusion Criteria:

* Non-ambulant people and people with a recent (e.g. within 6 months) cardiovascular disease event (e.g. stroke, myocardial infarction) or cardiac surgery,
* people with insulin-controlled diabetes mellitus or with coexisting skin conditions, leg ulcers, vasculitis or deep venous occlusion (as these may affect their cardiovascular function),
* pregnant women,
* people who require major surgery (which will prevent them of taking part in the study)
* people who following referral to the smoking cessation services, are advised that Nicotine Replacement Therapy is not appropriate for them,
* people who are currently using e-cigarettes on a daily basis, or currently undertaking an attempt within a smoking cessation service,
* people who are judged to be unable or are unwilling to give informed consent.

The study team will assess prospective participants and will not include in the study those who appear too frail or have health problems (e.g. dementia, Alzheimer's etc.) that might prevent them of giving a conscious, informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Intervention effect on Flow-mediated dilatation (FMD) assessed via ultrasound (%FMD). | 6 months following quit day.
  Macro-vascular function assessment.

SECONDARY OUTCOMES:
Intervention effect on Flow-mediated dilatation assessed via ultrasound (%FMD). | 3 days and 3 months following quit day.
  Macro-vascular function assessment.
Intervention effect on Laser Doppler Flowmetry (Perfusion Units). | 3 days, 3 months and 6 months following quit day.
  Micro-vascular function assessment.
Intervention effect on Mean Arterial Pressure. | 3 and 6 months following quit day.
  Mean arterial pressure assessment.
Intervention effect on Total Cholesterol/LDL ratio. | 3 and 6 months following quit day.
  Finger prick test (Total Cholesterol/LDL).
Intervention effect on Cardiovascular disease risk-reduction (Q-Risk assessment score). | 3 and 6 months following quit day.
  Q-risk assessment.
Patient experiences' assessment (Interview). | 3 months following quit day.
  Interview assessments of patient experiences.
Health Economics (Cost Utility Analysis). | 6 months following quit day.
  Health economic assessment of the intervention.
Carbon Monoxide assessment | 3 days, 3 months and 6 months following quit day.
  Carbon Monoxide assessment
Mean Arterial Pressure | 3 days, 3 months and 6 months following quit day.
  Mean arterial pressure assessments

OTHER OUTCOMES:
Physical activity assessment | 3 months and 6 months following quit day.
  Short Form (SF)- International Physical Activity Questionnaire (IPAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Markos Klonizakis, DPhil, Principal Investigator — Reader (Clinical Physiology)
Locations (1):
- Sheffield Hallam University, Sheffield, Yorkshire, United Kingdom

REFERENCES:
- [Derived] Klonizakis M, Gumber A, McIntosh E, Brose LS. Medium- and longer-term cardiovascular effects of e-cigarettes in adults making a stop-smoking attempt: a randomized controlled trial. BMC Med. 2022 Aug 16;20(1):276. doi: 10.1186/s12916-022-02451-9. PMID 35971150
- [Derived] Jones G, McIntosh E, Brose LS, Klonizakis M. Participant Experiences of a Quit Smoking Attempt Through Either Nicotine Replacement Therapy (NRT) Methods or the Use of an E-cigarette. J Addict Med. 2022 May-Jun 01;16(3):272-277. doi: 10.1097/ADM.0000000000000881. PMID 34128486
- [Derived] Klonizakis M, Crank H, Gumber A, Brose LS. Smokers making a quit attempt using e-cigarettes with or without nicotine or prescription nicotine replacement therapy: Impact on cardiovascular function (ISME-NRT) - a study protocol. BMC Public Health. 2017 Apr 4;17(1):293. doi: 10.1186/s12889-017-4206-y. PMID 28376818